CLINICAL TRIAL: NCT03979261
Title: Gender Study on Predisposition to Infectious Endocarditis
Brief Title: Predisposition to Infectious Endocarditis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-58; 2018-A02503-52 (Registry Identifier: APHM)
Record Dates: First submitted 2019-06-06; First posted 2019-06-07 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sex ratio evaluation: Valvular surgery is performed in 30-40% of cases. The Cardiology and Cardiac Surgery De la Timone services 1000 patients as part of their valvulopathy and 450 benefit from cardiac surgery. On the other hand, transcriptomic analysis by microarray will only be done on 40 patients because the analysis costs 150 € / patients.
  Interventions: Diagnostic Test: evolution of sex ratio according to age

INTERVENTIONS:
Diagnostic Test: evolution of sex ratio according to age — Histological study of the collected valves to study the differences according to the sex of the inflammatory reaction and the cellular type found.

SUMMARY:
To evaluate the gender-related elements, a first step will be to analyze the impact of sex ratio on different parameters such as age in endocarditis and the type of underlying valvulopathy and other associated comorbidities.

DETAILED DESCRIPTION:
Numerous epidemiological studies have made it possible to highlight the impact of the genus on the occurrence and natural evolution of numerous valvulopathies. Severe valve leakage occurs more frequently in men. This association is also observed in patients with aortic bicuspid infarction where infective endocarditis (IE) is 3 times more common in men with a sex ratio of 9 to 2 to 1. Male sex is also a risk factor of AEs in the admission score used in initial patient management used to stratify the risk of AE and start probabilistic antibiotic therapy. Several hypotheses were evoked and none made it possible to understand the impact of sex on the risk of IE. The transcriptome study of IE patients revealed 2 potential biomarkers. S100A11 (S100 calcium binding protein A11) is a diagnostic marker and AQP9 (Aquaporin 9 gene) a poor prognostic factor in patients with AE. Coxiella burnetii AE is more common and more severe in humans. A study in the C57 / BL6 mouse demonstrated the role of 17 beta-estradiol in decreasing bacterial load and granuloma formation in female mice. The hypothesis formulated is that sex hormones play a role in the natural history of IS. This hypothesis was confirmed at the transcriptome level in mice and allowed to identify transcriptomic signatures according to sex; male mice with a more marked inflammatory response to C. burnetii. In order to evaluate the gender-related elements, an initial work will be to analyze the impact of sex ratio on different parameters such as age in endocarditis and the type of underlying valvulopathy and other associated comorbidities.

The second part of the project will study (i) the transcriptional profile of the native valves removed in patients with endocarditis-free valvulopathy in male and female subjects (ii) the transcriptional profile of native valves removed during endocarditis in matching sex underlying valvulopathy and microorganism. This will evaluate a possible difference in susceptibility to endocardial fixation. (iii) the transcriptional profile of PBMCs (circulating mononuclear cells) in this same patient, which will make it possible to study the transcriptional profile of the circulating genes and to evaluate the possible difference in predisposition to endocardial fixation.

Finally, the third part will focus on the histological analysis of the valves collected to study the differences between man and woman (local inflammatory reaction, cell type found).

ELIGIBILITY:
Inclusion Criteria:

* Patient with infectious endocarditis
* Patient with valvulopathy or infective endocarditis requiring cardiac surgery as part of routine care.
* Major patient
* Patient informed of the study and having expressed no opposition to participate in the study.
* Patient affiliated to a social security scheme.

Exclusion Criteria:

* Minor patient
* Pregnant or nursing patient.
* Patient deprived of liberty or under judicial decision.
* Major patient under tutorship or curatorship.
* Patient not agreeing to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with valvulopathy or infective endocarditis requiring cardiac surgery as part of routine care.
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of sex ratio as a function of age and underlying pathologies (comorbidities and valvulopathies) | 36 months

SECONDARY OUTCOMES:
transcriptional profile by microarray | 36 months
  rate of indigenous valves removed in patients with valvulopathy without endocarditis by gender

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — AP HM
Locations (1):
- Laboratoires d'immunologie et d'infectiologie, Marseille, Cedex 5, France